CLINICAL TRIAL: NCT05095207
Title: A Multicenter, Phase IB/II Study of Abemaciclib in Combination With Bicalutamide for Androgen Receptor-positive, HER2-negative Metastatic Breast Cancer
Brief Title: Abemaciclib in Combination With Bicalutamide for Androgen Receptor-positive, HER2-negative Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amy Tiersten, Professor - Hematology Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 21-0699
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Metastasis
Keywords: Breast Cancer; Androgen Receptor-positive; HER2 negative; Abemaciclib; Bicalutamide
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — abemaciclib; bicalutamide

STUDY DESIGN:
Intervention Model Description: For the Phase 1 portion of the trial Bayesian optimal interval (BOIN) design is being used. a minimum of 3 and a maximum of 12 patients enrolled to determine RP2D. The 3-9 patients evaluated at the RP2D of the Phase I part of the trial will be enrolled and included in the Phase II part of the trial. If 2 or fewer among 12 patients in the first stage of Phase II have disease control, the trial will stop. However, if at least 3 have disease control in the first stage, then an additional 33 patients will be enrolled in the second stage, for a total of 46 patients. If among the 46 patients, 12 or fewer achieved complete response, partial response or stable disease, the treatment regimen under investigation in this trial will be rejected; or if at least 13 out of the 46 patients respond, the treatment regimen will be considered worthy of further study. The total sample size for Phase I and II portions combined is a minimum of 3 and a maximum of 60.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Androgen Receptor-positive, HER2-negative Metastatic Breast Cancer (Experimental): Abemaciclib in Combination with Bicalutamide
  Interventions: Drug: Abemaciclib; Drug: Bicalutamide

INTERVENTIONS:
Drug: Abemaciclib — 100 mg orally twice daily, day 1 to 28. If no toxicity in cycle 1 for the first 3 patients, increase dose to 150mg orally twice daily day 1-28 and enroll 3 patients. If excessive toxicity experienced at 100mg orally twice daily dose, decrease dose to 50mg orally twice daily day 1-28.
Drug: Bicalutamide — 150 mg orally daily, day 1 to 28.

SUMMARY:
This is an open label multicenter, Phase IB/II Study of Abemaciclib in Combination with Bicalutamide for Androgen Receptor-positive, HER2-negative Metastatic Breast Cancer

DETAILED DESCRIPTION:
This is an open label multicenter, Phase IB/II Study of Abemaciclib in Combination with Bicalutamide for Androgen Receptor-positive, HER2-negative Metastatic Breast Cancer About 54-60 patients will be enrolled over the course of 36 months. Patients will be treated until disease progression.

Study regimen is Abemaciclib with Bicalutamide

Primary objective is to determine the dose-limiting toxicity (DLT) and recommended phase II dose for abemaciclib when administered in combination with bicalutamide and to determine the efficacy of the treatment secondary objective is to determine the safety and tolerability along with progression free survival.

Given the suggestive pre-clinical data and the unique properties of abemaciclib, the researchers believe that abemaciclib is an ideal partner for bicalutamide in treatment of AR+ metastatic breast cancer. The study team hypothesize that the combination will demonstrate a further improved clinical benefit rate than either agent alone, including in those patients who have already been treated with prior endocrine therapies. Additionally, the study team believe that the convenience of an all-oral, continuous daily dosing schedule and the favorable side effect profile of both therapies with minimal overlapping or serious toxicities further supports this investigation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses

  * If a patient declines to participate in any voluntary exploratory research and/or genetic component of the study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study
* Women aged at least 18 years
* The patient has a biopsy-confirmed diagnosis of recurrent, unresectable, locally advanced, or metastatic HER2neu-negative breast cancer (including bone-only metastatic disease) o The patient must have had biopsy confirmation of a metastatic site (with appropriate ER/PR/HER2neu IHC staining)

  o The patient has measurable or evaluable disease as evidenced on pre-treatment baseline CT chest, abdomen, and pelvis with bone scan OR PET/CT
* The patient has AR+ breast cancer (defined as > or equal to 1% staining on immunohistochemistry of metastatic breast cancer specimen)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
* If the patient has ER+ or PR+ (>1% on IHC) metastatic breast cancer:

  o patient must have had 1 prior line of endocrine therapy in the metastatic setting
  * prior CDK4/6 inhibitor exposure allowed (abemaciclib. palbociclib, or ribociclib)
  * no more than 2 prior line of cytotoxic chemotherapy in the metastatic setting allowed
* If the patient has ER-,PR-, HER2- metastatic breast cancer ("triple-negative"):

  o The patient may have had up to 4 prior lines of chemotherapy in the metastatic setting and at least 1 prior line of chemotherapy in the metastatic setting
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy).
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
* Post-menopausal status or receiving ovarian ablation with a GnRH agonist such as goserelin or leuprolide. Postmenopausal status is defined by any one of the following criteria:

  * Prior bilateral oophorectomy.
  * Age ≥ 60 years.
  * Age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, or ovarian suppression) and FSH, LH, and estradiol in the postmenopausal range per local normal.

If the patient does not meet criteria for postmenopausal status but is receiving ovarian ablation therapy with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin or leuprolide, the patient is eligible for the study, provided that the GnRH agonist is started at least 2 weeks prior to C1D1 of study therapy.

- Negative serum pregnancy test within 7 days prior to starting treatment

• Women of child-bearing potential and men must agree to use a highly effective method of contraception prior to study entry, for the duration of study participation, and for 3 weeks following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately, as cases of pregnancy that occur during maternal exposures to abemaciclib should be reported. If a patient or spouse/partner is determined to be pregnant following abemaciclib initiation, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are to be collected for regulatory reporting and drug safety evaluation.

Note: Recommended methods of birth control are: The consistent use of an intrauterine device (IUD), Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam), Sexual abstinence (no sexual intercourse) or Sterilization.

Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 90 days after completion of therapy.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* Treatment with any of the following:

  1. Any investigational agents or study drugs from a previous clinical study within 28 days of the first dose of study treatment
  2. Any other chemotherapy, immunotherapy or anticancer agents within 21 days of the first dose of study treatment
  3. Any prior exposure to anti-androgen therapy (bicalutamide, abiraterone, and/or enzalutamide)
* Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
* Spinal cord compression, leptomeningeal carcinomatosis, or brain metastases - unless asymptomatic, treated and stable and not requiring steroids for at least 2 weeks prior to start of study treatment
* Concurrent use of endocrine therapy (tamoxifen, anastrozole, letrozole, exemestane, oral contraceptive pills)
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 consecutive electrocardiograms (ECGs)
  2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block)
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, abnormalities in serum electrolytes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
  4. Personal history of syncope of cardiovascular etiology, ventricular arrhythmia (of pathologic origin including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
  5. Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA Grade 2 or greater
  6. Uncontrolled hypotension - Systolic BP <90mmHg and/or diastolic BP <50mmHg
  7. Left ventricular ejection fraction (LVEF) below lower limit of normal for site
* Prior history of DVT/PE or embolic stroke, unless currently on therapeutic anticoagulation
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  1. Absolute neutrophil count < 1.5 x 109/L
  2. Platelet count < 100 x 109/L
  3. Hemoglobin < 8 g/L (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.)
  4. Alanine aminotransferase > 3 times the upper limit of normal (ULN)
  5. Aspartate aminotransferase > 3 times ULN
  6. Total bilirubin > 1.5 times ULN (patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted)
  7. Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN
  8. Proteinuria 3+ on dipstick analysis or >500mg/24 hours
  9. Sodium or potassium outside normal reference range for site
* Liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis. Patients who are hepatitis B Core antibody IgG positive are allowed to participate if taking and compliant with daily oral hepatitis B prophylactic medications
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 89% or less at rest on room air
* Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption abemaciclib or bicalutamide
* Patients with an active bleeding diathesis
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* History of hypersensitivity or allergic reaction to abemaciclib or bicalutamide, or drugs with a similar chemical structure or class
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Co-administration with CYP3A4 inducers (e.g., phenytoin, rifampin, carbamazepine, St John's Wort, bosentan, efavirenz, etravirine, modafinil, and nafcillin), CYP3A4 inhibitors (e.g., clarithromycin, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, verapamil, and voriconazole), and CYP3A4 substrates (e.g., alfentanil, cyclosporine, dihydroergotamine, ergotamine, everolimus, fentanyl, pimozide, quinidine, sirolimus and tacrolimus). See Appendix C for complete list.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Female patients who are pregnant or breast feeding/lactating, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a method of contraception.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All Female All Male
Enrollment: 42 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Dose-Limiting Toxicity (DLT) and Recommended Phase II Dose (RP2D) | 12 weeks
  For the Phase 1 portion of the trial Bayesian optimal interval (BOIN) design is being used. a minimum of 3 and a maximum of 12 patients enrolled to determine the dose-limiting toxicity (DLT) and will be the recommended phase II dose (RP2D).
  • A DLT will be defined as:
  * Grade 3 or 4 non-hematologic toxicity
  * Grade 3 neutropenia lasting greater than 21 days
  * Grade 3 or 4 neutropenia with neutropenic fever
  * Grade 4 hematologic toxicity events experienced within the first 4 weeks (1 cycle) of study treatment.
  These will be assessed via National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v.5.0 toxicity criteria. The DLT period will be the first cycle (28 days) of therapy.

SECONDARY OUTCOMES:
Frequency of Adverse Events (AE) | 12 weeks
  The frequency and percentage of AE associated with abemaciclib in combination with bicalutamide by the type, severity (as graded by the NCI CTCAE v.5.0), and relationship to study medications.
Disease Control Rate (DCR) | 12 weeks
  Disease Control Rate (DCR) is defined as the percentage of patients whose cancer shrinks or remains stable over the duration of the study. This will be measured as the sum of complete response (CR), partial response (PR), and stable disease (SD) for greater than or equal to 24 weeks.
  CR: Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
  PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
  PD: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai - West, New York, New York
  - Dubin breast Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. To achieve aims in the approved proposal. Information will be made once available